CLINICAL TRIAL: NCT03939091
Title: Ultrasonographic Versus Renographic Parameters in Prediction of Early Success After Pyeloplasty in Children. A Prospective Study.
Brief Title: Ultrasonographic Versus Renographic Parameters in Prediction of Early Success After Pyeloplasty in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohamed Abdelazeem, Principal Investigator, Mansoura University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Renogram.US.Pyeloplasty
Record Dates: First submitted 2019-04-23; First posted 2019-05-06 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-04

CONDITIONS: Pyeloplasty; Pediatrics; Renogram; Ultrasonography
Keywords: Ultrasonography; Pyeloplasty; Renogram; Follow up
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ultrasonography (Other): Renal Ultrasonography
  Interventions: Diagnostic Test: Ultrasonography

INTERVENTIONS:
Diagnostic Test: Ultrasonography — Renal Ultrasonography

SUMMARY:
To study the predictive value of ultrasonographic (USG) parameters in the form of anteroposterior diameter , calyceal dilatation , calyx-to-parenchyma ratio , renal length , renal width , pelvis-to-cortex ratio (PCR) and parenchymal thickness versus renographic parameters in the form of T1/2 , differential renal function (DRF) and Tissue tracer transit (TTT) for early detection of children at risk of recurrent obstruction post unilateral pyeloplasty.

ELIGIBILITY:
Inclusion Criteria:

* patients who will be scedueled for pyeloplasty

Exclusion Criteria:

* bilateral pathology
* Pelvi-ureteric junction obstruction (PUJO) in a solitary kidney
* other associated anomalies

Ages: 6 Months to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
evaluate predictive value of ultrasonographic parameters for early detection of recurrent obstruction | 30 months
  assessed by Diuretic scintigraphy (T1/2) as the time it takes for the activity in the kidney to decrease to 50% of its maximum value measured in minutes
evaluate predictive value of ultrasonographic parameters for early detection of decrease renal function | 30 months
  assessed by Diuretic scintigraphy differential renal function (DRF) measured in millilitres/minute

CONTACTS AND LOCATIONS:
Locations (1):
- Urology and nephrology center, Al Mansurah, Outside U.S./Canada, Egypt

IPD SHARING:
Plan to Share IPD: No